CLINICAL TRIAL: NCT03616665
Title: Feasibility and Effectiveness of a Personalized Inpatient Program Tailored for Persistent Depressive Disorder With Childhood Maltreatment and Comorbidity: Personalized Cognitive Behavioral Analysis System of Psychotherapy
Brief Title: Feasibility and Effectiveness of a Personalized Inpatient Program for Persistent Depressive Disorder
Acronym: PePsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Philipps University Marburg (Other)
Collaborators: Schön Klinik Bad Arolsen (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018_14k
Record Dates: First submitted 2018-06-28; First posted 2018-08-06 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: Persistent Depressive Disorder
Keywords: persistent depressive disorder; psychotherapy; cognitive behavioral therapy; inpatient treatment; childhood maltreatment; treatment-resistance; clinical effectiveness; personalized psychotherapy; comorbidity; cognitive behavioral analysis system of psychotherapy; online aftercare
MeSH Terms: interventions — Pharmaceutical Preparations

STUDY DESIGN:
Intervention Model Description: In the proposed prospective, mono-site, evaluator-blinded study, 100 PDD patients will be included. The study addresses the primary research question: Is the six-week inpatient CBASPersonalized-treatment effective in PDD? It is hypothesized that six weeks after randomization, CBASPersonalized will evoke significant reduction in depressive symptomatology. In addition, feasibility will be examined and differential indication by moderator, process and long-term analyses will be investigated. A follow-up survey six months after end of treatment will provide important results on long-term treatment outcome.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CBASPersonalized (Other): Within the psychotherapy CBASPersonalized, the original specific six interpersonal CBASP strategies are augmented with intrapersonal evidence-based strategies. According to the frequently diagnosed comorbid disorders of PDD the following modules have been added: a) treatment of anxiety disorders and treatment of traumatic experiences, b) regulating intensive emotions, c) coping with resistant problems like pain, and d) relapse prevention. In addition, therapists adjust their strategies and therapeutic relationship according to the impairment in personality functioning and maladaptive personality traits of the patient.
  Interventions: Other: CBASPersonalized

INTERVENTIONS:
Other: CBASPersonalized — In addition to CBASPersonalized patients will receive algorithm-based pharmacotherapy in compliance with current national and international guidelines for depression treatment and according to clinical expert supervision. Of note, the intake of the medication is documented and taken into account in the analyses.
  After completion of the six-week inpatient treatment, patients will be offered the six-to-twelve-week blended-online-aftercare CBASPersonalized@home.
  Patients are allowed to attend additional inpatient groups like creative and sports therapy. The participation in these groups is documented.
  Other Names: Drug

SUMMARY:
The major objective of this study is to evaluate a new conceptualized personalized concept of Cognitive Behavioral Analysis System of Psychotherapy (CBASPersonalized) in the treatment of patients with persistent depressive disorder (PDD), childhood maltreatment and a high rate of comorbidity. Patients receive a two-phase-treatment-program (six-weeks inpatient-treatment and six-to-twelve-weeks blended-online-aftercare) in combination with standardized pharmacotherapy in a routine clinical inpatient setting. This study addresses the primary research question: Is an intensive six-week inpatient CBASPersonalized treatment feasible and effective in a clinical sample of PDD patients? In addition, moderator, process and long-term analyses will be conducted for differential insights.

DETAILED DESCRIPTION:
Background: Persistent depressive disorder (PDD) is a prevalent disabling disorder. Given its high degree of treatment-resistance (TR), comorbidity, and suicidality, this patient group constitutes a massive health problem. The Cognitive Behavioral Analysis System of Psychotherapy (CBASP) was specifically developed for the outpatient treatment of PDD showing superiority to active control groups in some studies. However, non-remission and relapse rates of CBASP are relatively high, which might be caused by the fact that within the original CBASP-concept the frequent comorbid disorders are not sufficiently addressed. Thus, an optimized personalized short and intensive CBASP-concept (CBASPersonalized) was established including the interpersonal CBASP-strategies while adding evidence-based intrapersonal strategies being tailored to the specific comorbid problems. In this study, the investigators will evaluate the feasibility and effectiveness of CBASPersonalized. Patients will receive a six-week inpatient treatment followed by a six-to-twelve-week blended-online-aftercare (CBASPersonalized@home) in combination with standardized pharmacotherapy in a routine clinical inpatient setting.

Methods: In the proposed prospective, mono-site study, 100 PDD patients with childhood maltreatment will be included. The study addresses the primary research question: Is an intensive six-week inpatient CBASPersonalized treatment feasible and effective in a clinical sample of PDD patients? It is hypothesized that six weeks after admission, CBASPersonalized will evoke significant reduction in depressive symptomatology (according to the 24-item version of the Hamilton Rating Scale of Depression, HRSD). The feasibility (acceptance and subjective experience) is assessed on the basis of the dropout rate and a self-assessed questionnaire, which measures satisfaction with and subjective effectiveness of the specific treatment components.

In addition, moderator, process and long-term analyses will be conducted for differential insights. Primary and secondary outcome will be analyzed using analysis of covariance (ANCOVA) controlling for pre-treatment scores. Moderator and process analyses will be performed using multiple regression and linear mixed models.

As a specific secondary research question, we will examine the associations between childhood maltreatment (CM), depression severity, and potential psychological mechanisms of this associations (emotion regulation, self-compassion, empathic distress, interpersonal problems) at the beginning of treatment. In addition, we will explore which changes in the potential psychological mechanisms are particularly closely related to changes in depressive symptoms.

As another additional research question, we will examine the associations between the state-like therapeutic alliance, trait-like alliance, and depression severity. We want to explore these associations as a possible effect mechanism and specify a possible transfer to CBASP specific mechanisms of actions.

Finally, the analyses of the outcomes at the end of the six-to-twelve week blended online-aftercare and the follow-up survey 6 months after end of treatment will provide important results on the blended after-care program as well as longterm treatment outcome. Of note, we will evaluate the online continuation treatment CBASPersonalized@home regarding feasibility. Therefore, patients' expectations towards the intervention, their adherence (completed modules and exercises), acceptance and satisfaction with the intervention as well as the perceived fit and perceived effectiveness and usability of the intervention will be analyzed. Depression severity at the beginning of CBASPersonalized@home, expectations, satisfaction and therapeutic alliance will be analyzed as possible predictors of adherence. A possible relationship between changes in depressive symptoms in the course of the continuation treatment and adherence will be explored.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of persistent depressive disorder (PDD) according to DSM-5
* Experiences of childhood maltreatment (>Cut-off criteria in one of 5 scales of the Childhood Trauma Screener (CTS))
* Sufficient German language skills
* Have read and signed an informed consent form

Exclusion Criteria:

* Life-time diagnosis of an schizophrenia or schizophrenic spectrum disorder according to DSM-5
* Life-time diagnosis of a schizoid, schizotypal or antisocial personality disorder according to DSM-5
* Consumption of legal (e.g. alcohol) or illegal substances during the inpatient stay

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Hamilton Rating Scale of Depression, 24-item version (HRSD-24) | The primary outcome is given by the post value (week six: end of inpatient treatment) in the HRSD24.
  The change in HDRS-24 item score (Hamilton, 1960; Williams, 1988) from baseline to 6 weeks after study start will be the primary endpoint. The HRSD-24 is a semi-structured interview which is used to measure the severity of all symptom domains of depression as described by the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) over a period of the last 7 days. It shows good psychometric properties. The HRSD-24 will be conducted by blind study raters at every time point. Raters evaluate symptom severity on a scale from 0 to 2 or 0 - 3 or 0 - 4 for each item, with higher number indicating higher symptom severity. The total score ranges from 0 to 75 with higher values indicating higher depression severity.

SECONDARY OUTCOMES:
Beck Depression Inventory-II (BDI-II) | Baseline, 2, 4, 6, 8, 9, 14, and 37 weeks after study start
  Self-report instrument to assess the severity of depression on 21 items, each symptom represents one item with responses from 0 (symptom absent) to 4 (symptom present). The total score ranges from 0 to 63 with higher values indicating more severe depressive symptoms.
Montgomery Asberg Depression Rating Scale (MADRS) | Baseline, 2, 4, 6, 14, and 37 weeks after study start
  Observer-report instrument to assess the severity of depression (symptom areas: apparent sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, suicidal thoughts) on a 7-point Likert scale with 6 representing highest severity. In the applied MADRS+ version, three items assessing helplessness, hopelessness and worthlessness are added. Hence, the total score of MADRS+ ranges from 0 - 71 with higher values indicating more severe depression.
Brief Symptom Inventory (BSI) | Baseline, 6, 14, and 37 weeks after study start
  Self-report questionnaire to assess general psychopathological symptom severity in nine different symptom dimensions (somatization, obsessive-compulsive, interpersonal sensitivity, depression, anxiety, hostility, phobic anxiety, paranoid ideation, psychoticism, general severity score) on a scale from 0 to 4 with 4 representing more severe symptoms. A global indicator is the General Severity Index (GSI) which will be used as a total score here. The GSI is given by the mean of all subscales and ranges from 0 (low general symptom severity) to 4 (high severity).
Patient Health Questionnaire (PHQ) | Baseline, 6, 14, and 37 weeks after study start
  Self-report questionnaire for the assessment of various mental health conditions (factors are somatic, anxiety and depression symptom scales), responses are given on a scale from 0 to 2 (with 2 representing higher symptom severity)
Inventory of Personality Organization (IPO-16) | Baseline, 6, 14, and 37 weeks after study start
  Self-report measure for the assessment of personality dysfunction in three domains (identity, defense, reality-testing)
revised Impact of Event Scale (IES-R) | Baseline, 6, 14, and 37 weeks after study start
  self-report of post-traumatic stress symptoms with the three subdomains intrusions, avoidance and over-arousal; a scoring scheme with intervals of 0 (not at all), 1 (rarely), 3 (sometimes), and 5 (often) is used to reflect frequency of symptoms over the past week. Subscales are analyzed by summing up all responses of items that belong to one subscale. Intrusion and hyperarousal range between 0 - 35 and avoidance ranges between 0 - 40, with higher values indicating more severe intrusion/ hyperarousal/ avoidance.
Social Support Questionnaire F-SozU | Baseline, 6, 14, and 37 weeks after study start
  self-report to assess perceived social support on the four scales emotional and practical support, social integration, and social stress. Additional scales are reciprocity, availability of a trusted person, satisfaction with social support. Contains 54 items; responses are given on a 5-point Likert scale. Patients indicate their level of agreement with a presented statement from 0 (totally disagreed) to 4 (totally agreed). The total range is from 0 to 216 with higher values representing higher perceived and received social support.
Depressive Expectations Scale (DES) | Baseline, 6, 14, and 37 weeks after study start
  self-report to assess intensity of dysfunctional expectations (regarding social rejection/ support, mood regulation and the ability to perform). The DES consists of 25 items. Responses are given on a 5-point Likert-scale where patients express their agreement with a given statement (1= I don't agree to 5= I agree). The total score varies between 0 and 125 with higher values indicating higher intensity of dysfunctional expectations.
Difficulties in Emotion Regulation Scale (DERS) | Baseline, 6, 14, and 37 weeks after study start
  self-report to assess the flexibility and adaptiveness of emotion regulation. The DERS consists of 36 items. Responses are given on a 5-point Likert-scale where patients indicate how often the following statements apply to them (1= almost never (0-10%) to 5= almost always (91-100%). The total score varies between 0 and 180 with higher scores suggesting greater problems with emotion regulation.
revised Adult Attachment Scale (AAS-R) | Baseline, 6, 14, and 37 weeks after study start
  self-report to assess individual's attachment style on the subscales closeness, trust and anxiety; on a scale from 1 (not at all true) to 5 (very true). There are 15 items in total with 5 belonging to each subscale. Higher values reflect higher comfort with closeness or depending on others or concern about abandonment.
Self-Compassion Scale-Short Form (SCS-SF) | Baseline, 6, 14, and 37 weeks after study start
  self-report to assess six components of self-compassion (self-kindness, self-judgement, common humanity, isolation, mindfulness, over-identification). Response format ist a 5-point Likert-type scale ranging from 1 (almost never) to 5 (almost always). Total scores can range between 0 and 60 with higher values representing higher levels of self-compassion.
Impact Message Inventory (IMI-R) | Baseline, 6, 14, and 37 weeks after study start
  observer-rated questionnaire designed to measure distinctive internal reactions, referred to as impact messages, that interactants experience to the full range of interpersonal behaviours indexed along the circumplex of the interpersonal circle with the 2 dimensions dominance-submissiveness and friendliness-hostility. Messages are rated on a scale from 0 (not at all) to 4 (very much). The total score of each subscale is considered for analysis.
Measure of Disorders of Capacity as defined by the International Classification of Functioning (MINI-ICF) | Baseline, 6, 14, and 37 weeks after study start
  observer-rated questionnaire to measure quality of life and functioning, framed as skill deficits in 12 areas (e.g. skill to adapt to rules and routines, professional and non-professional skills, assertiveness, endurance etc.) Skill deficits are assessed using a response scale from 0 (no skill deficits) to 4 (complete absence of skill)
Health-related quality of life (EQ-5D-5L) | Baseline, 6, 14, and 37 weeks after study start
  self-rated questionnaire to measure health-related quality of life. Health is assessed using 5 dimensions: mobility, self-care, usual activities, pain/ discomfort, anxiety/ depression. For each dimensions, participants can select one option out of 5 that describes them best.
Euthymia Scale (ES) | Baseline, 6, 14, and 37 weeks after study start
  self-rated questionnaire to assess euthymia. It contains 10 items which assess factors of general mood, energy and coping with stressors. Responses are given by selecting (True/ False) for a specific statement. The total range of the ES is from 0 to 10 with 10 indicating higher prevalence of euthymia.
Working Alliance Inventory (WAI-SR) | T0 for WAI-e; WAI-C and WAI-T at 1, 2, 3, 4, 5, 6; WAI-C at 13, and 37 weeks after study start
  Self-rated questionnaire administered to patients (WAI-C) and therapists (WAI-T) to assess the quality of the working alliance based on Bordin's pan theoretical concept via 3 subscales (12 items each): a)goals: agreement about the goals of therapy; b)tasks: agreement about the tasks of therapy, c)bond: bond between therapist and patient. Responses are given on a 7-point Likert scale (1= totally disagree, 7= totally agree). Mean scores are analysed for all 3 subscales and on an overall level, with higher values indicating higher satisfaction with the therapeutic alliance.
  Patient expectations of alliance are assessed via an adapted form of the WAI-SR (WAI-expected; WAI-e) prior to the start of therapy at an initial assessment (T0). The instructions are altered by adding the following sentence: "Since you have not yet received any therapy through this study, we ask you to think about what you expect from the therapy in answering the following questions."
Global Assessment of Functioning (GAF) | Baseline, 6, 14, and 37 weeks after study start
  observer-rated questionnaire to measure functioning in 9 descriptors (work, law, social (family and friends), judgement, thinking, mood, anxiety, hallucinations, suicidal ideation). Each descriptor has a 9-point range from 0 (most severe) to 90 (least severe)
PATHEV (Patient Therapy Expectation and Evaluation questionnaire) | The PATHEV is administered at an initial assessment (T0), prior to the start of therapy.
  The PATHEV is a questionnaire measuring patient expectations on three scales: (1) hope of improvement, (2) fear of change, and (3) suitability (Schulte, 2005). It consists of 11 items and is rated on a 5-point Likert scale. The instrument has shown acceptable to good reliability (Cronbachs Alpha 0.73- 0.89). Construct validity of the scales has been demonstrated via three studies.
WAI-e (WAI-expected) | Assessed prior to the start of therapy at an initial assessment (T0).
  Patient expectations of alliance were assessed by an adapted form of the WAI-SR (WAI-expected, WAI-e).
  The instructions were altered by adding the following sentence: "Since you have not yet received any therapy through this study, we ask you to think about what you expect from the therapy in answering the following questions."
Interpersonal Reactivity Index (IRI) | Baseline, 6, 14, and 37 weeks after study start
  To assess dispositional empathic traits, a shortened and validated German version of the interpersonal reactivity index (IRI) self-report survey is used (Davis, 1980; German Version: Paulus, 2009). The questionnaire measures the four domains (1.) perspective-taking, (2.) empathic concern, (3.) personal distress, and (4.) fantasy with four items per subscale.
Evaluation of CBASPersonalized inpatient treatment | At the end of the inpatient treatment, 6 weeks after study start
  A self-constructed questionnaire concerning patients' fit, acceptance and satisfaction is used to evaluate the CBASPersonalized inpatient treatment. Patients are asked to evaluate the therapy components individually according to these three criteria. All items were answered on a 6-level Likert scale.

OTHER OUTCOMES:
Moderator variable: Childhood Trauma Questionnaire (CTQ-SF) | baseline
  Childhood maltreatment will be assessed using the short version of the Childhood Trauma Questionnaire (CTQ-SF) measuring the five subscales emotional abuse, emotional neglect, sexual abuse, physical abuse, and physical neglect. 12 additional Items are added to the original questionnaire to measure experiences of inconsistency and the age (or age-span) at which the participant was exposed to childhood maltreatment.
Process variable: Inventory of Interpersonal Problems (IIP) | Baseline, 6, 14 and 37 weeks after study start
  It will be examined whether the effectiveness of CBASPersonalized can be explained by an improvement of interpersonal problems in CBASP. The IIP is a self-rated questionnaire to assess a variety of interpersonal problems.
General Self-Efficacy Scale (GSE; Jerusalem & Schwarzer, 1999) | Baseline, 6, 14 and 37 weeks after study start
  Patients' perceived general self-efficacy is assessed using the 10-items version of the SWE. Items are rated on a 4-piont Likert-scale. Total score can be interpreted using age and gender specific standard scores.
Videoconference and Telepresence Scale (VTS; Bouchard & Robillard, 2000) | 9 and 12 weeks after study start
  The questionnaire measures naturalness of a videoconference therapy by the percentage of agreement (0-100%) with eight statements. The original version shows preliminary validation (α =.84). For this study, the English version was translated into German.
Session Evaluation Questionnaire (SEQ; Stiles & Snow, 1984) | 9 and 12 weeks after study start
  This 21 items questionnaire examines the participant's satisfaction with a therapeutic session and can be divided into four subscales (depth, smoothness, positivity, arousal). Items are rated on a seven-point Likert scale ranging from for example 1 to 7. The questionnaire shows high internal consistency.
System Usability Scale (SUS; Brooke, 1986) | 9 and 12 weeks after study start
  This self-report-questionnaire is a "quick and dirty" method which outlines the usability of a system in percentage terms. The German version of the 10-item-inventory was adapted to the videoconference setting of the study as recommended by the author. A five point Likert scale ranging from 1 to 5 is used to rate the items. The high economy and validity of the SUS justify its use in the present study (Brooke, 1986).
Client Satisfaction Questionnaire adapted to Internet-based interventions (CSQ-I; Boß et al., 2016) | 9, 12 and 14 weeks after study start
  The CSQ-I consists of 8 items measuring global satisfaction with online interventions. Items are rated on a 4-point Likert-scale. Good construct validity and high internal consistency has been shown in one study.
Working Alliance Inventory for guided Internet Interventions (WAI-I; Penedo et al., 2019) | 9, 12 and 14 weeks after study start
  Therapeutic alliance in the guided online aftercare is measured using the WAI-I, which is an adapted version of the WAI-SR focusing on guided internet interventions. Twelve items rated on are 5-piont Likert-scale are divided into three subscales (bond, goal, task). The questionnaire which is shows adequate internal consistency and external validity in one study so far.
Evaluation of CBASPersonalized@home online continuation treatment | At the end of the online continuation treatment, 14 weeks after study start
  A self-constructed questionnaire with 16 items concerning patients' acceptance (4 items; e.g. "I find the use of CBASPersonalized@home following the inpatient treatment useful"), fit (3 items; e.g. "I have the feeling that CBASPersonalized@home was exactly right for me and my problems") and subjective effectiveness (9 items; e.g. " Through CBASPersonalized@home I have a better understanding of the views and feelings of other people.") is used to evaluate the online continuation program CBASPersonalized@home. All items were answered on a 6-level Likert scale.
  Patients' usage behavior is assessed with five additional items which are answered categorially.

CONTACTS AND LOCATIONS:
Overall Officials: Eva-Lotta Brakemeier, Prof. Dr., Study Chair — University Greifswald and Philipps University Marburg; Jörg-Tobias Hof, Principal Investigator — Schön Klinik Bad Arolsen (study site)
Locations (2):
- Germany (2):
  - Schoen Klinik Bad Arolsen, Bad Arolsen, Hesse
  - Philipps University Marburg, Faculty psychology, department clinical psychology, Marburg, Hesse

IPD SHARING:
Plan to Share IPD: Yes
Individual patient data will be shared with researchers providing a clinical relevant and methodological sound proposal.
Supporting Information: SAP, ICF, Analytic Code
Time Frame: These above mentioned proposals should be submitted within 48 months following first publication of the main results of this trial.